CLINICAL TRIAL: NCT05253885
Title: Smartphone Addiction in Relation to Trunk Position Sense, Fatigue and Insomnia in Adolescences
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Shaimaa Shawky Muhammad, Principal investigator, October 6 University
Other Study IDs: smartphone003
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Adolescent Behavior; Smartphone Addiction
MeSH Terms: conditions — Adolescent Behavior; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smartphone addiction group
  Interventions: Device: Smartphone use

INTERVENTIONS:
Device: Smartphone use — * Smartphone addiction scale (short version) higher than 33
  * Smartphone users of 4-5 inches screen size smartphones, weighing 140-160 grams and dimensions less than 159*79*9 mm.

SUMMARY:
The aim of the study is to evaluate the relationship between smartphone addiction and trunk position sense, insomnia and fatigue in adolescents. Sample size will be determined after a pilot study conducted on a small sample of adolescents. Digital goniometer will be used to evaluate trunk position sense, insomnia severity index will be used to evaluate insomnia severity and fatigue will be measured by fatigue severity scale.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with age between 17 and 18 years old.
* BMI between 16.4 and 24.8 kg/m2
* Smartphone addiction scale (short version) higher than 33
* Smartphone users of 4-5 inches screen size smartphones, weighing 140-160 grams and dimensions less than 159*79*9 mm.

Exclusion Criteria:

* Visual or hearing defects.
* Congenital abnormalities.
* Neurological abnormalities
* Musculoskeletal abnormalities

Ages: 17 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: - Adolescents with age between 17 and 18 years old with Smartphone addiction scale (short version) higher than 33
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-25 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Trunk position sense | Single measurement (instant measure)
  Digital goniometer will be used to determine trunk position sense. Procedure will be performed with open-closed eye positions with a trunk flexion and trunk lateral bending right/left without any verbal feedback from the examiner. It will be measured in terms of repositioning error angle (the difference between reached and targeted angles).
Insomnia severity index | Single measurement (instant measure)
  Insomnia severity will be assessed by insomnia severity index. It contains 7 items and each participant will read each statement and check a number from 0 to 4. respondents use five point LIKERT scale to rate each item (example: 0= no problem, 4= very severe problems).
Fatigue severity scale | Single measurement (instant measure)
  Arabic version of fatigue severity scale will be used to determine fatigue level. It contains 9 items as each participant will be asked to read each statement and circle a number from 1(completely disagree) to 7 "completely agree"/

CONTACTS AND LOCATIONS:
Overall Officials: Elham E Salem, Professor of Physical Therapy, Study Chair — Cairo University; Walaa A Abdelnabie, Professor of Physical Therapy, Study Director — Cairo University
Locations (1):
- October 6 University hospital, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided